CLINICAL TRIAL: NCT03556059
Title: Procedure Selection in Obesity and Metabolic Surgery Based on the Edmonton Obesity Staging System (EOSS) - a Nationwide German Register-based Cohort Study (StuDoQ MBE)
Brief Title: Procedure Selection in Obesity and Metabolic Surgery Based on EOSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sana Klinikum Offenbach (Other)
Collaborators: Deutsche Gesellschaft für Allgemein- und Viszeralchirurgie (Other)
Responsible Party: Principal Investigator, Sonja Chiappetta, MD, Senior consultant, Principal Investigator, MD, Sana Klinikum Offenbach
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FF 83_2/2015
Record Dates: First submitted 2018-05-18; First posted 2018-06-14 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Postoperative Complications
Keywords: EOSS; Obesity and metabolic surgery; postoperative outcome; procedure selection
MeSH Terms: conditions — Postoperative Complications; Obesity

STUDY DESIGN:
Intervention Model Description: A cohort of all patients who underwent obesity and metabolic surgery in Germany will be analyzed in relation to preoperative complications
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RNYGB (Active Comparator): The role of EOSS for the surgical intervention: Roux-en-Y gastric bypass for severe obesity
  Interventions: Other: Role of EOSS
- Sleeve (Active Comparator): The role of EOSS for the surgical intervention: Sleeve Gastrectomy for severe obesity
  Interventions: Other: Role of EOSS
- MGB/OAGB (Active Comparator): The role of EOSS for the surgical intervention: Mini/One anastomosis gastric bypass for severe obesity
  Interventions: Other: Role of EOSS

INTERVENTIONS:
Other: Role of EOSS — The Edmonton Obesity Staging System (EOSS) is a more comprehensive measure of obesity-related diseases and predictor of mortality than body mass index (BMI) or waist circumference. Its application for the selection of obese patients for obesity surgery has been suggested. This study evaluates the role of the Edmonton Obesity Staging System (EOSS) in predicting postoperative outcome (next to the Clavien Dindo Classification) and 30-day mortality after metabolic surgery.

SUMMARY:
The Edmonton Obesity Staging System (EOSS) is a more comprehensive measure of obesity-related diseases and predictor of mortality than BMI or waist circumference. EOSS is also important in predicting post - operative outcome and 30-day mortality after metabolic surgery.

The aim of this study is to determine whether EOSS could be an indicator for procedure selection in obesity and metabolic surgery.

DETAILED DESCRIPTION:
All patients in Germany, who underwent Sleeve Gastrectomy, Roux-en Y Gastric Bypass and Mini/One anastomosis Gastric Bypass as a primary procedure for severe obesity, are prospectively registered in the German register StuDoQ MBE.

Preoperative EOSS by Sharma et al. will be applied to all patients, who were operated between Februar 2015 and July 2017 by two different evaluators. Data collection will include the following: gender, age, body mass index, mobility, comorbidities, ASA score (American Society of Anesthesiologists score) perioperative complications next to Clavien Dindo, readmission rates and 30 - day mortality. Follow-up will be investigated in all patients up to 1 month after surgery.

Complications, readmission rates and 30 day mortality will be investigated in relation to EOSS and the surgical procedure performed, to determine whether EOSS could be an indicator for procedure selection in obesity and metabolic surgery.

ELIGIBILITY:
Inclusion Criteria:

Sleeve for severe obesity RNYGB for severe obesity MGB/OAGB for severe obesity

-

Exclusion Criteria:

* previous obesity surgery
* previous surgery of the upper gastrointestinal tract in anamnesis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9437 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
postoperative complications | 30 days after surgery
  postoperative outcome after surgery next to the Clavien Dindo Classification

SECONDARY OUTCOMES:
postoperative complications related to surgical procedure | 30 days after surgery
  postoperative complications related to surgical procedure
postoperative complications related to Edmonton Obesity Staging System | 30 days after surgery
  postoperative complications related to Edmonton Obesity Staging System
ASA related to Edmonton Obesity Staging System | prior to surgery
  ASA related to Edmonton Obesity Staging System
Edmonton Obesity Staging System related to length of postoperative stay | 30 days after surgery
  Edmonton Obesity Staging System related to length of postoperative stay
Edmonton Obesity Staging System related to readmission | 30 days after surgery
  Edmonton Obesity Staging System related to readmission
Edmonton Obesity Staging System related gender | 30 days after surgery
  Edmonton Obesity Staging System related gender
Edmonton Obesity Staging System related to surgical procedure | 30 days after surgery
  Edmonton Obesity Staging System related to surgical procedure
postoperative complications related to ASA | 30 days after surgery
  postoperative complications related to ASA
postoperative complications related to gender | 30 days after surgery
  postoperative complications related to gender
age related to postoperative complications | 30 days after surgery
  age related to postoperative complications
Body Mass Index related to postoperative complications | 30 days after surgery
  Body Mass Index related to postoperative complications
Edmonton Obesity Staging System related to age | 30 days after surgery
  Edmonton Obesity Staging System related to age
Edmonton Obesity Staging System related to Body Mass Index | 30 days after surgery
  Edmonton Obesity Staging System related to Body Mass Index

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Weiner, Prof., Study Director — Sana Klinikum Offenbach
Locations (1):
- Sana Klinikum Offenbach, Offenbach, Germany

IPD SHARING:
Plan to Share IPD: No
Anonymous data will be published in a peer-reviewed journal.

REFERENCES:
- [Result] Sharma AM, Kushner RF. A proposed clinical staging system for obesity. Int J Obes (Lond). 2009 Mar;33(3):289-95. doi: 10.1038/ijo.2009.2. Epub 2009 Feb 3. PMID 19188927
- [Result] Kuk JL, Ardern CI, Church TS, Sharma AM, Padwal R, Sui X, Blair SN. Edmonton Obesity Staging System: association with weight history and mortality risk. Appl Physiol Nutr Metab. 2011 Aug;36(4):570-6. doi: 10.1139/h11-058. Epub 2011 Aug 14. PMID 21838602
- [Result] Padwal RS, Pajewski NM, Allison DB, Sharma AM. Using the Edmonton obesity staging system to predict mortality in a population-representative cohort of people with overweight and obesity. CMAJ. 2011 Oct 4;183(14):E1059-66. doi: 10.1503/cmaj.110387. Epub 2011 Aug 15. PMID 21844111
- [Result] Gill RS, Karmali S, Sharma AM. The potential role of the Edmonton obesity staging system in determining indications for bariatric surgery. Obes Surg. 2011 Dec;21(12):1947-9. doi: 10.1007/s11695-011-0533-8. No abstract available. PMID 22002510
- [Result] Chiappetta S, Stier C, Squillante S, Theodoridou S, Weiner RA. The importance of the Edmonton Obesity Staging System in predicting postoperative outcome and 30-day mortality after metabolic surgery. Surg Obes Relat Dis. 2016 Dec;12(10):1847-1855. doi: 10.1016/j.soard.2016.02.042. Epub 2016 Mar 2. PMID 27317606
- [Derived] Chiappetta S, Stier C, Weiner RA; members of StuDoQ|MBE of Deutsche Gesellschaft fur Allgemein- und Viszeralchirurgie/StuDoQ. The Edmonton Obesity Staging System Predicts Perioperative Complications and Procedure Choice in Obesity and Metabolic Surgery-a German Nationwide Register-Based Cohort Study (StuDoQ|MBE). Obes Surg. 2019 Dec;29(12):3791-3799. doi: 10.1007/s11695-019-04015-y. PMID 31264178